CLINICAL TRIAL: NCT05881551
Title: Clinical Pain Assessment Via Force Measurement Using the eEgg in the Setting of Routine Elective Lumbar Facet Joint Blocks (SMeEgg): a Prospective, Randomized, Two-arm Pilot Study.
Brief Title: Pain Assessment Via Force Measurement Using eEgg After Blockade of the Lumbar Facet Joints
Acronym: SMeEgg
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Witten/Herdecke (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: SMeEgg
Record Dates: First submitted 2023-04-21; First posted 2023-05-31 (Actual); Last update posted 2024-03-25 (Actual); Status verified 2024-03

CONDITIONS: Pain Measurement
Keywords: pain measurement; blockade of the lumbar facet joints; peri-interventional; grip strenth; chronic pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- eEgg-Arm (Experimental): Within the 24h interval, pain assessment is performed hourly using the NRS (during the day) and the eEgg (preferably at hourly intervals throughout the day). If necessary, additional measurements can be taken with the eEgg.
  Interventions: Device: eEgg
- NRS-Arm (Other): Patients are asked to document their current pain at hourly intervals for 24 hours (starting from the end of the intervention) according to the usual clinical routine. The first measurement is taken before the intervention.
  Interventions: Other: NRS

INTERVENTIONS:
Device: eEgg — In the eEgg-Arm, patients are given the eEgg immediately before the intervention to familiarize themselves with this method. Here, the patient is asked to press the device with maximum force for five seconds, which would correspond to an NRS value of 10, and to press the eEgg only with half force, which corresponds to an NRS value of 5. Following the instruction, the current pain score present is recorded and documented using the NRS and the eEgg. The same procedure takes place at the end of the 24h observation interval when the eEgg is returned. Within the 24h interval, pain assessment is performed hourly using the NRS (during the day) and the eEgg (preferably at hourly intervals throughout the day). If necessary, additional measurements can be taken with the eEgg.
  Arms: eEgg-Arm
Other: NRS — Patients record their pain on the numeric rating scale (NRS) within the 24-hour interval. An interval from 0 to 10 is given (0 = no pain, 10 = most pain imaginable).
  Arms: NRS-Arm

SUMMARY:
The emotion Egg, or "eEgg" for short, is a sample series of a device for testing a new pain measurement method that is not yet on the market. The aim is to investigate whether the trial device and the eEgg method (eEgg plus software) are suitable for supporting, improving or even replacing the communication between doctor and patient, which still takes place via the numerical rating scale (NRS) and the pain diary. Issues of acceptability in comparison to the pain diary and the NRS are to be considered. Measurements should be recorded in real time; no orientation to the previous value is possible for the patient.

ELIGIBILITY:
Inclusion Criteria:

* Elective interventional blockade of lumbar facet joints due to lumbar facet osteoarthritis
* Chronic pain (>3 months, most severe pain on motion in the last three months ≥3 (NRS))
* Age ≥18 years
* Legal capacity
* Proficiency in the German language
* Presence of a written informed consent from the patient
* Inpatient pain patient

Exclusion Criteria:

* Participation in other interventional trials
* Individuals who have a dependent/employee relationship with the sponsor or investigator
* Cognitive impairment that could affect the use of the eEgg
* Impaired fist closure and/or reduction of gross strength in the hand area
* mono- or poly-neuropathy in the hand area
* Allergy to plastics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2023-05-22 (Actual); Primary Completion 2024-01-08 (Actual); Study Completion 2024-01-08 (Actual)

PRIMARY OUTCOMES:
Comparison of the expressions of pain ratings in eEgg-Arm and in NRS-Arm | immediately after blockade for 24 hours
  For the analysis of pain ratings using eEgg versus NRS (numerical rating scale, values 0-10 [0=no pain - 10=the most severe pain imaginable]), functional data analysis methods are used to account for the longitudinal structure of the data. In a first step, the pain rating measurements are transformed into continuous smooth curves based on B-spline basis functions. Then, a functional principal component analysis based on the fitted curves is performed to analyze the temporal variation.
  Suitable statistical measures (median/mean, quartiles/standard deviation, etc.) are used to describe the primary target variable. If necessary, a suitable statistical test follows, such as the Mann-Whitney U test for the group comparison.

SECONDARY OUTCOMES:
Comparison of the expressions of the pain ratings within eEgg-Arm | immediately after blockade for 24 hours
  For the analysis of pain ratings using eEgg versus NRS (numerical rating scale, values 0-10 [0=no pain - 10=the most severe pain imaginable]), functional data analysis methods are used to account for the longitudinal structure of the data. In a first step, the pain rating measurements are transformed into continuous smooth curves based on B-spline basis functions. Then, a functional principal component analysis based on the fitted curves is performed to analyze the temporal variation.
Comparison of pain rating by NRS from eEgg-Arm with pain rating by NRS from NRS-Arm | immediately after blockade for 24 hours
  NRS: numerical rating scale, values 0-10 [0=no pain - 10=the most severe pain imaginable]
  The secondary outcome measures are evaluated using appropriate statistical measures of location (median/mean, quartiles/standard deviation, frequencies/percentages, etc.). If necessary, appropriate statistical significance tests are performed to compare measurements between the two randomization groups (e.g. for continuous data Mann-Whitney U test, e.g. for categorical data Fisher's exact test or Chi² test) or within the groups (e.g. for continuous data sign test, e.g. for categorical data McNemar test).
Number of measurements with the eEgg during the night | immediately after blockade for 24 hours
  The secondary outcome measures are evaluated using appropriate statistical measures of location (median/mean, quartiles/standard deviation, frequencies/percentages, etc.). If necessary, appropriate statistical significance tests are performed to compare measurements between the two randomization groups (e.g. for continuous data Mann-Whitney U test, e.g. for categorical data Fisher's exact test or Chi² test) or within the groups (e.g. for continuous data sign test, e.g. for categorical data McNemar test).
Comparison of the standardization values in the eEgg group at the beginning of the study | before the blockade
  The secondary outcome measures are evaluated using appropriate statistical measures of location (median/mean, quartiles/standard deviation, frequencies/percentages, etc.). If necessary, appropriate statistical significance tests are performed to compare measurements between the two randomization groups (e.g. for continuous data Mann-Whitney U test, e.g. for categorical data Fisher's exact test or Chi² test) or within the groups (e.g. for continuous data sign test, e.g. for categorical data McNemar test).
Comparison of the standardization values in the eEgg group at the end of the study | 24 hours after the blockade
  The secondary outcome measures are evaluated using appropriate statistical measures of location (median/mean, quartiles/standard deviation, frequencies/percentages, etc.). If necessary, appropriate statistical significance tests are performed to compare measurements between the two randomization groups (e.g. for continuous data Mann-Whitney U test, e.g. for categorical data Fisher's exact test or Chi² test) or within the groups (e.g. for continuous data sign test, e.g. for categorical data McNemar test).
Difference in pain sensation (NRS) due to the different local anesthetics | immediately after blockade for 24 hours
  NRS: numerical rating scale, values 0-10 [0=no pain - 10=the most severe pain imaginable]
  The secondary outcome measures are evaluated using appropriate statistical measures of location (median/mean, quartiles/standard deviation, frequencies/percentages, etc.). If necessary, appropriate statistical significance tests are performed to compare measurements between the two randomization groups (e.g. for continuous data Mann-Whitney U test, e.g. for categorical data Fisher's exact test or Chi² test) or within the groups (e.g. for continuous data sign test, e.g. for categorical data McNemar test).
Questionnaire evaluation on the handling of the eEgg | 24 hours after the blockade
  The secondary outcome measures are evaluated using appropriate statistical measures of location (median/mean, quartiles/standard deviation, frequencies/percentages, etc.). If necessary, appropriate statistical significance tests are performed to compare measurements between the two randomization groups (e.g. for continuous data Mann-Whitney U test, e.g. for categorical data Fisher's exact test or Chi² test) or within the groups (e.g. for continuous data sign test, e.g. for categorical data McNemar test).

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Cegla, Dr., Principal Investigator — Helios University Hospital Wuppertal
Locations (1):
- Helios Universitätsklinikum Wuppertal, Wuppertal, Germany